CLINICAL TRIAL: NCT00451399
Title: Efficacy of Lifestyle Interventions and Metformin for the Treatment of Antipsychotic-Induced Weight Gain: a Randomized Double-Blind Placebo- Controlled Comparison
Brief Title: Efficacy of Lifestyle Interventions and Metformin for the Treatment of Antipsychotic-Induced Weight Gain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central South University (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Jzhao
Expanded Access: Available
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Weight Gain
Keywords: Weight gain; antipsychotic; lifestyle interventions; metformin; antipsychotic-induced weight gain.
MeSH Terms: conditions — Weight Gain | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: metformin
Behavioral: lifestyle intervention

SUMMARY:
Lifestyle intervention and certain medications have been shown to be effective for antipsychotic-induced weight gain, but no controlled studies have compared psychological and pharmacological therapies. We conducted a randomized, placebo-controlled study to test the efficacy of lifestyle intervention and metformin alone and in combination for antipsychotic-induced weight gain.

DETAILED DESCRIPTION:
The study was designed as a double-blind randomized controlled trial, with research assessors and patients intended to be blind to the intervention status. The staff members performing the assessment were not involved in implementing any aspect of the intervention.128 patients were randomized to one of four 12-week individual treatments: metformin (750mg/day), placebo, lifestyle intervention plus metformin (750mg/day) or lifestyle intervention plus placebo. Medications were provided in double-blind fashion.The assessments include body weight, body mass index, waist circumference, fasting glucose, fasting insulin and insulin resistance index.

ELIGIBILITY:
Inclusion Criteria:

* All participants met the Diagnostic and Statistical Manual of Mental Disorder-Fourth Edition (DSM-Ⅳ) criteria for schizophrenia27.
* Participants were required to get weight gain more than 10% of their predrug body weight during less than 12 months of treatment with a targeted antipsychotic agent- clozapine, olanzapine, risperidone or sulpiride.
* The duration of illness for all participants was less than 12 months.
* Participants could be taking only one antipsychotic, whose dose had not changed by changed by more than 25% over the past 3 months.
* All patients were stable outpatient.
* The total score of Positive and Negative Syndrome Scale (PANSS) for all patients could be ≤60.
* All participants were ensured that they could be carefully taken care of by one of their parents or guardians during the trial.

Exclusion Criteria:

* Participants were excluded from the study if they had evidence of liver or renal diseases, pregnant or lactating women, cardiovascular diseases, hypertension or diabetes mellitus, specific systemic diseases, or conditions that limited their ability to perform the lifestyle modifications, such as arthritis, pulmonary diseases, neurological or dietary restrictions.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128
Dates: Start 2004-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
body weight, body mass index, waist circumference, fasting glucose, fasting insulin, insulin resistance index

CONTACTS AND LOCATIONS:
Overall Officials: Jingping Zhao, MD, Study Director — Second Xiangya Hospital of Central South University
Locations (1):
- Institute of Mental Health of The Second Xiangya Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Derived] Kang D, Jing Z, Li R, Hei G, Shao T, Li L, Sun M, Yang Y, Wang Y, Wang X, Long Y, Huang X, Wu R. Effect of Betahistine and Metformin on Antipsychotic-Induced Weight Gain: An Analysis of Two Clinical Trials. Front Psychiatry. 2018 Nov 27;9:620. doi: 10.3389/fpsyt.2018.00620. eCollection 2018. PMID 30542300
- [Derived] Wu RR, Zhao JP, Jin H, Shao P, Fang MS, Guo XF, He YQ, Liu YJ, Chen JD, Li LH. Lifestyle intervention and metformin for treatment of antipsychotic-induced weight gain: a randomized controlled trial. JAMA. 2008 Jan 9;299(2):185-93. doi: 10.1001/jama.2007.56-b. PMID 18182600